CLINICAL TRIAL: NCT03802669
Title: Molecular Assessment of Oral Mutans Streptococcus Isolated From Patients With Different Age and Caries Activity Via Selective Media and Protein Pattern.
Brief Title: Molecular Assessment of Oral Mutans Streptococcus Isolated From Different Patients
Status: Completed | Type: Observational
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Naglaa Ibrahim Ezz, Lecturer of pediatric dentistry department, faculty of dentistry, October University for Modern Sciences and Arts
Other Study IDs: ETH10
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Dental Caries
Keywords: human saliva; mutans streptococcus; PCR; caries activity
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- caries free children aged between 3-6
  Interventions: Other: oral mutans streptococcus
- caries active children aged between 3-6
  Interventions: Other: oral mutans streptococcus
- caries free children aged between 6-12
  Interventions: Other: oral mutans streptococcus
- caries active children aged between 6-12
  Interventions: Other: oral mutans streptococcus
- caries free adult aged between 18-25
  Interventions: Other: oral mutans streptococcus
- caries active adult aged between 18-25
  Interventions: Other: oral mutans streptococcus

INTERVENTIONS:
Other: oral mutans streptococcus — quantitative assessment of mutans streptococcus of each group by using PCR and protein pattern

SUMMARY:
90 saliva samples will be isolated from patient who possess different ages and caries activity, attending outpatient clinic of October University of Modern Sciences and Arts. Then the determination of the best selective media for mutans streptococcus isolated from saliva and authenticate the MS via PCR technique.

ELIGIBILITY:
Inclusion Criteria:

* healthy participant

Exclusion Criteria:

* participant received antimicrobial therapy in previous month.
* participant who taking xylitol chewing gum or undergo fluoride therapy.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients attending out patient clinic of October University for Modern Sciences and Arts.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
oral mutans streptococcus screening | immediately
  screening of oral mutans streptococcus of each group to determine the differences

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa Ezzeldin, lecturer, Principal Investigator — October University for Modern Sciences and Arts
Locations (1):
- October University of Modern Sciences and Arts, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No